CLINICAL TRIAL: NCT05554341
Title: Nilotinib and Paclitaxel in Patients With Prior Taxane-Treated Solid Tumors: A ComboMATCH Treatment Trial
Brief Title: Testing the Use of Nilotinib and Paclitaxel as a Treatment for Patients With Prior Taxane Treatment, A ComboMATCH Treatment Trial
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-07264; NCI-2022-07264 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY191-E4 (Other: ECOG-ACRIN Cancer Research Group); EAY191-E4 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2022-09-22; First posted 2022-09-26 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Malignant Solid Neoplasm; Refractory Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; nilotinib; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (nilotinib hydrochloride monohydrate, paclitaxel) (Experimental): Patients receive nilotinib hydrochloride monohydrate PO BID on days 1-28 and paclitaxel IV over 1 hour on days 1, 8, and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT or MRI throughout the study. Patients also undergo collection of blood samples and tumor biopsy on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Nilotinib Hydrochloride Monohydrate; Drug: Paclitaxel

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Nilotinib Hydrochloride Monohydrate — Given PO
  Other Names: AMN 107; AMN-107; AMN107; Nilotinib Monohydrochloride Monohydrate; Tasigna
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat

SUMMARY:
This phase II ComboMATCH treatment trial evaluates nilotinib with paclitaxel for the treatment of patients with solid cancers that are growing, spreading, or getting worse (progressive) and that have previously been treated with taxane therapies. Nilotinib is in a class of medications called kinase inhibitors. It works by binding to and blocking the action of a protein called ABL, which signals tumor cells to multiply. This helps slow or stop the proliferation of tumor cells. Paclitaxel is a drug that blocks cell growth by stopping cell division and it may kill tumor cells. Giving nilotinib with paclitaxel may be effective at treating patients with progressive solid cancers that have previously been treated with taxane therapies.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with taxane-refractory advanced malignancies who have objective responses (OR) to treatment with nilotinib hydrochloride monohydrate (nilotinib) and paclitaxel.

SECONDARY OBJECTIVE:

I. Collect tissue and provide it to the ComboMATCH registration protocol to assess concordance between the diagnostic tumor mutation profile generated by the designated laboratories, the pre-treatment biopsy mutation profile, and the pre-treatment circulating tumor deoxyribonucleic acid (ctDNA) mutation profile from plasma, as described in ComboMATCH registration protocol. For this treatment substudy, the outcome objective will be to report the proportion of cases providing sufficient tissue for that integrated scientific activity in the ComboMATCH registration protocol.

EXPLORATORY OBJECTIVES:

I. To evaluate progression free survival (PFS) at 6 months on study agents. II. To identify genomic and transcriptomic determinants of response and resistance in tumor biopsy specimens and cell-free deoxyribonucleic acid (DNA).

OUTLINE:

Patients receive nilotinib hydrochloride monohydrate orally (PO) twice daily (BID) on days 1-28 and paclitaxel intravenously (IV) over 1 hour on days 1, 8, and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) or magnetic resonance imaging (MRI) throughout the study. Patients also undergo collection of blood samples and tumor biopsy on study.

After completion of study treatment, patients are followed until disease progression, and for survival for 3 years from registration.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be enrolled on the ComboMATCH registration protocol (EAY191) at the time of registration to the EAY191-E4 study
* Patient must be >= 18 years of age
* Patient must not have any of the following mutations (as determined by the ComboMATCH registration protocol), which are known to confer sensitivity or resistance to nilotinib monotherapy:

  * KIT: W557R, V559D, V559A, L576P, and K642E
  * PDGFR-alpha: D842V
* Patient must have disease that can be safely biopsied and agree to a pre-treatment biopsy or have archival tissue available from within 12 months prior to the date of registration on the ComboMATCH registration trial (EAY191)

  * NOTE: The current actionable mutation of interest (aMOI)/actionable alteration list for this treatment trial can be found on the Cancer Trials Support Unit (CTSU) website
  * NOTE: Novel/dynamic aMOI can be submitted for review per the process described in the ComboMATCH registration protocol
* Patient must be willing to provide blood samples for research purposes
* Patient must have had at least one prior line of therapy in the metastatic setting
* Patient must have previously undergone taxane therapy (in the metastatic setting)

  * Patients who previously responded to prior taxane therapy must have received their last dose of taxane therapy within 6 months prior to EAY191-E4 registration and have had no other intervening treatment prior to EAY191-E4 registration
  * Patients who did not respond to prior taxane therapy are eligible regardless of the time elapsed since the prior taxane therapy or any other intervening therapies
* Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Patient must not have had platinum-resistant epithelial serous ovarian cancer
* Patients must not have neuropathy >= grade 2 within 14 days of registration/randomization
* Patient must have documented QT interval with Fridericia's correction (QTcF) of =< 450 msec within 8 days prior to EAY191-E4 registration. Patients with a QTcF interval of >= 450 msec at registration or patients with congenital long QT syndrome are not eligible
* Patient must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used

  * All patients of childbearing potential must have a blood test or urine study within 14 days prior to registration to rule out pregnancy
  * A patient of childbearing potential is defined as anyone, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Patient must not expect to conceive or father children by using accepted and effective method(s) of contraception or by abstaining from sexual intercourse for the duration of their participation in the study and for at least 3 months after the last dose of study drug
* Patients must have progressive disease
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (with the exception of those with Gilbert syndrome, who must have total bilirubin =< 3 x institutional ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 institutional upper limit of normal; < 5.0 x ULN in patients with liver metastases
* Creatinine clearance > 60 mL/min/1.73 m^2 for patients with creatinine levels > 1.5 mg/dL
* Patient must have the ability to swallow medications
* Patient must have completed any prior therapy ≥ 4 weeks or ≥ 5 half-lives of the prior agent (whichever is shorter) prior to enrollment on protocol. Prior definitive radiation should have been completed ≥ 4 weeks prior to enrollment; prior palliative radiation should have been completed ≥ 2 weeks prior to enrollment. Patients must be ≥ 2 weeks since any investigational agent administered as part of a phase 0 study (where a sub-therapeutic dose of drug is administered) and should have recovered to grade 1 or baseline from any toxicities
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression for ≥ 1 month after treatment of the brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Best objective response | Up to 3 years
  Evaluated using Response Evaluation Criteria in Solid Tumors version 1.1. 90% two-sided confidence intervals will be used for reporting estimated rates.
Progression free survival | From registration to documented disease progression or death from any cause, assessed up to 3 years
  Distribution will be estimated using the method of Kaplan and Meier.
Overall survival | From registration to death from any cause, assessed up to 3 years
  Distribution will be estimated using the method of Kaplan and Meier.
Incidence of adverse events | Up to 3 years
  Will be determined using the National Cancer Institute's Common Terminology Criteria for Adverse Events. Exact binomial confidence intervals will be used for adverse event rates.

SECONDARY OUTCOMES:
Concordance of diagnostic tumor mutation profile, pre-treatment tumor biopsy mutation profile, and pre-treatment circulating tumor deoxyribonucleic acid (ctDNA) profile | Up to 3 years
  Whole-exome sequencing, ribonucleic acid sequencing, and ctDNA sequencing will be performed on mandatory tissue biopsies and/or blood specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Shin, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (126):
- United States (126):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Kingman Regional Medical Center, Kingman, Arizona
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mount Sinai Hospital, New York, New York
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - M D Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Valley Medical Center, Renton, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT05554341/ICF_000.pdf